CLINICAL TRIAL: NCT01517321
Title: MK-0431/ONO-5435 Phase III Clinical Trial-Rapid-acting Insulin Secretagogue Add-on Study in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: MSD K.K. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5435-17; Japic CTI-111668 (Registry Identifier: Japan Pharmaceutical Information Center)
Record Dates: First submitted 2011-11-02; First posted 2012-01-25 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- E (Experimental)
  Interventions: Drug: MK-0431/ONO-5435
- P (Placebo Comparator)
  Interventions: Drug: Placebo, MK-0431/ONO-5435

INTERVENTIONS:
Drug: MK-0431/ONO-5435 — Double-blind period (12 wk); 50 mg QD. The double-blind period will be followed by a 40 week open label extension period where MK-0431/ONO-5435 could be titrated from 50 mg to 100 mg QD.
  Arms: E
Drug: Placebo, MK-0431/ONO-5435 — Double-blind period (12 wks); placebo QD. The double-blind period will be followed by a 40 wk open label extension period where MK-0431/ONO-5435 could be titrated from 50 mg to 100 mg QD.
  Arms: P

SUMMARY:
This Phase III clinical trial will examine the safety, tolerability, and efficacy of the addition of MK-0431/ONO-5435 to Japanese patients with Type 2 Diabetes mellitus who have inadequate glycemic control on diet/exercise therapy and rapid-acting insulin secretagogue monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on diet/exercise therapy and rapid-acting insulin secretagogue monotherapy

Exclusion Criteria:

* Patients with Type 1 Diabetes Mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Incidences of adverse experiences and change in vital sign, safety lab etc. as parameters of safety and tolerability | 12 weeks and 52 weeks

SECONDARY OUTCOMES:
HbA1c | 12 weeks
2-hour postmeal glucose | 12 weeks
Fasting plasma glucose | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akiteru Seki, Study Chair — First Division Clinical Development Planning 1
Locations (6):
- Japan (6):
  - Chugoku Region Clinical Site, Chugoku
  - Chubu Region Clinical Site, Chūbu
  - Kanto Region Clinical Site, Kanto
  - Kinki Region Clinical Site, Kinki
  - Kyusyu Region Clinical Site, Kyusyu
  - Tohoku Region Clinical Site, Tōhoku